CLINICAL TRIAL: NCT05421455
Title: Surgical Intervention Versus Biologics Treatment for Symptomatic Stricturing Crohn's Disease (SIBTC): an Open-label, Single-center, Randomized Controlled Trial
Brief Title: Surgery Versus Biologics for Stricturing CD--a RCT
Acronym: SIBTC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhu Weiming (Other)
Responsible Party: Sponsor-Investigator, Zhu Weiming, chief of general surgery, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: jinlingH20220609
Record Dates: First submitted 2022-06-09; First posted 2022-06-16 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biologic group (Other): treat paticipants with up to 2 biologics
  Interventions: Drug: Group A
- Surgery group (Other): treat paticipants with surgery
  Interventions: Procedure: Group B

INTERVENTIONS:
Drug: Group A — treat participants with biologics
  Arms: Biologic group
Procedure: Group B — treat participants with surgery
  Arms: Surgery group

SUMMARY:
The management of stricturing Crohn's disease (CD) remains challenging. Although surgical resection may be the final way to solve it, the efficacy of biologics for symptomatic CD associated strictures was acceptable. In clinical practice, the chioce of treatment is particularly difficult. Therefore, a clinical trial of biologics versus surgery is needed to assess which one is prefered.

ELIGIBILITY:
Inclusion Criteria:

1. with intestinal obstructive symptoms;
2. confirmed intestinal strictures;
3. traditional drugs failed to induce remission;
4. envidence of active bowel inflammation;
5. inappropriate for EBD;
6. acquirement of written informed consent of participant;

Exclusion Criteria:

1. unsuccessful medical treatment of intestinal obstruction;
2. complete obstruction;
3. contraindication for biologics;
4. penetrating disease;
5. short smaal bowel;
6. suspicion of bowel tumor;
7. no confirmed strictures;
8. comitant severe disese of other system;
9. obstructive symptoms under over 2 targets of biologics;
10. successful treatment with traditional drugs;
11. participate other clinical research.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 138 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2025-06-09 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
clinical remmision rate within 1 year | within 1 year
  Crohn's disease activity index < 150

SECONDARY OUTCOMES:
inflammatory bowel disease score | within 1 and 5 year
  32-224；the higher the better
Crohn's disease obstructive score | within 1 and 5 year
  0-6； the higher the worse
endoscopic recurrence | within 1 and 5 year
  Rutgeert score >i2b (i0-i4); the higher the worse
medical cost | within 1 and 5 year
  cost for hospitalization
sugical recurrence | within 1 and 5 year
  disease recurrence that needs surgical resection
clinical remmision rate within 5 year | within 5 year
  CDAI>150

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Jinling hosptal,Medical School of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No